CLINICAL TRIAL: NCT03297801
Title: The Effects of Omega-3 Polyunsaturated Fatty Acids on the Infant Microbiome and Immunity
Brief Title: The Effects of Omega-3 PUFAs on the Infant Microbiome and Immunity
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Deanna Gibson, Associate Professor, University of British Columbia
Other Study IDs: H13-02523
Record Dates: First submitted 2017-09-25; First posted 2017-09-29 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Microbial Colonization; Infant Development
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fish oil group: Women who chose to supplement with fish oil, rich in omega-3 polyunsaturated fatty acids, during gestation or lactation.
  Interventions: Dietary Supplement: Fish oil supplements
- No fish oil group: Women who chose not to supplement with fish oil during gestation or lactation.

INTERVENTIONS:
Dietary Supplement: Fish oil supplements — Women who chose to supplement with fish oil during gestation or lactation.
  Groups: Fish oil group

SUMMARY:
Prenatal supplementation with fish oil, rich in omega-3 polyunsaturated fatty acids, is widely recommended in Canada. The aim of this observational, prospective cohort study is to determine the effects of maternal fish oil supplements on the development of their infants' gut microbiota and immunity.

DETAILED DESCRIPTION:
During infancy, the gastrointestinal tract is colonized with microbiota, a community of microorganisms, which play a significant role in the development, regulation, and maintenance of immune functions. Fish oil, rich in n-3 polyunsaturated fatty acids (PUFA), are thought to be anti-inflammatory and consequently may increase susceptibility to infection by hindering their body's ability to produce an adequate inflammatory response in defense against infectious disease. Currently, women in Canada are supplementing their diets with n-3 PUFA during gestation and lactation despite their being conflicting clinical evidence regarding the beneficial effects on infant development. It is currently unknown how maternal fish oil supplementation impacts the offspring's gut microbiota and immune functions. Considering that diet influences microbiota and maternal microbiota is passed from mother to infant, the investigators hypothesize that maternal fish oil supplementation will affect the participants' infant gut microbiota and immunity.

This study will evaluate the effects of postnatal n-3 PUFA supplementation in breast milk on the fecal microbiome in infants over a six-month period. The investigators will analyze the fecal microbiome of infants born to mothers in the fish oil and non-fish oil groups via next generation sequencing. As short-chain fatty acids (SCFA) are produced by gut bacteria and affect immunity, the investigators will analyze SCFA in stool through gas chromatography. Markers of inflammation like fecal calprotectin and sIgA in stool samples will also be identified.

ELIGIBILITY:
Inclusion Criteria:

* All mothers of infants in the Okanagan Valley are invited to participate in the study between the first day of delivery to until solid food is introduced into the infant's diet.
* Healthy, full-term infants, who are predominantly breastfed by mothers who are or are not supplementing with fish oil. Mothers must also be healthy, i.e., asymptomatic and with no clinical indication of disease.
* To remain within the inclusion criteria for this study, participants will be expected to be consistent (i.e. maintain the same type and amount of omega-3 PUFA intake or no intake) with whichever supplementation group they have decided to join for the entirety of the breast milk and infant stool donation period. In other words, the investigators will be asking the participants not to switch from one group to another which would happen by changing their omega-3 PUFA supplementation patterns.

Exclusion Criteria:

* Any infants who are ingesting juice or solid foods as part of their regular diet will be excluded from the study.
* Any infants who are clinically ill (fever, contagious diseases, or active diarrhea) will be excluded from the study.
* Any participants who decide to drastically change their omega-3 PUFA supplementation intake patterns (i.e. causing them to switch between study groups) will result in all subsequent samples to be excluded from the study.

Ages: 5 Days to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy women in the Okanagan Valley who predominantly breastfeed their healthy, full-term infants while self-administering fish oil supplements or not.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2014-01-22 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Changes in infant fecal microbiota of the two groups. | 6 months
  Fecal microbiota will be measured by examining microbial taxa from infant stool every month from birth until 6-months of age or until solids are introduced.

SECONDARY OUTCOMES:
Changes in infant short-chain fatty acid production of the two groups. | 6 months
  Changes in short-chain fatty acid production will be analyzed in infant stool through gas chromatography.
Changes in infant IgA in shed intestinal epithelial cells of the two groups. | 6 months
  We will examine the effects of fish oil on immunity by measuring fecal IgA concentrations using ELISA
Changes in infant cytokines in shed intestinal epithelial cells of the two groups. | 6 months
  We will examine the effects of fish oil on immunity by measuring fecal cytokines (TNF-a, IFN-y, IL-17) using real time PCR.
Compare occurrences of sickness and incidences of disease between the two groups. | 2 years
  Any incidences of disease in the infants will be closely monitored for the first 2 years of their lives.
Changes in breast milk IgA composition of the two groups. | 6 months
  Immune markers such as sIgA will be measured in breast milk using an addressable laser bead immunoassay (ALBIA)
Changes in breast milk cytokine composition of the two groups. | 6 months
  Immune markers such cytokines will be measured in breast milk using an addressable laser bead immunoassay (ALBIA)
Changes in breast milk lipid composition of the two groups. | 6 months
  Breast milk lipid concentrations will be analyzed using short-chain fatty acids

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L Gibson, Ph.D., Principal Investigator — University of British Columbia

IPD SHARING:
Plan to Share IPD: No
Infant stool microbial data will be made open access upon publishing.

REFERENCES:
- [Derived] Quin C, Estaki M, Vollman DM, Barnett JA, Gill SK, Gibson DL. Probiotic supplementation and associated infant gut microbiome and health: a cautionary retrospective clinical comparison. Sci Rep. 2018 May 29;8(1):8283. doi: 10.1038/s41598-018-26423-3. PMID 29844409